CLINICAL TRIAL: NCT04304859
Title: Brief Assessment of Impaired Cognition
Acronym: BASIC
Status: Completed | Type: Observational
Sponsor: Danish Dementia Research Centre (Network)
Responsible Party: Sponsor
Other Study IDs: NVD-2019-01; 1604063 (Other Grant/Funding Number: Danish Ministry of Health)
Record Dates: First submitted 2019-11-28; First posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Dementia
Keywords: validation; casefinding tool
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases referred from GP: BASIC (Brief Assessment of Impaired Cognition) MMSE (Mini Mental State Examination) Extensive diagnostic work-up including clinical interview, neurological and physical examination, laboratory screening tests, structural neuroimaging
  Interventions: Diagnostic Test: BASIC
- Healthy controls: Test performed:
  BASIC MMSE GDS-15 (Geriatric Depression Scale)
  Interventions: Diagnostic Test: BASIC

INTERVENTIONS:
Diagnostic Test: BASIC — Validation

SUMMARY:
The aim is to develop and validate a new brief and accurate case-finding instrument for dementia and cognitive impairment - BASIC

DETAILED DESCRIPTION:
The case-finding instrument consists of four components: a. patient-directed questions, b. supermarket fluency, c. category-cued Memory Test, d. informant-directed questions.

The data collection was carried out at five outpatient memory clinics in Denmark

ELIGIBILITY:
Inclusion Criteria:

* fluent in Danish

Exclusion Criteria:

* impaired eyesight or hearing

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Cases: Patients referred from GP for diagnostic evaluation Controls: Participating patients' relatives and volunteers from ongoing research projects at the involved memory clinics.
Sampling Method: Non-Probability Sample
Enrollment: 428 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Brief Assessment of Impaired Cognition (BASIC) | through study completion, an average of 1 year
  Dementia and cognitive impairment cutoff 20/21

CONTACTS AND LOCATIONS:
Overall Officials: Gunhild Waldemar, Study Director — Danish Dementia Research Centre
Locations (1):
- DDRC, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No